CLINICAL TRIAL: NCT01894061
Title: A Prospective Phase II Trial of NovoTTF-100A With Bevacizumab (Avastin) in Patients With Recurrent Glioblastoma
Brief Title: NovoTTF-100A With Bevacizumab (Avastin) in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3313
Record Dates: First submitted 2013-07-03; First posted 2013-07-09 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor; Bevacizumab-naive; NovoTTF-100A
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bevacizumab and NovoTTF-100A (Experimental): Bevacizumab will be administered intravenously on days 1 and 15 of each 28 day cycle.The dose of bevacizumab will be 10 mg/kg of actual body weight.
  Interventions: Biological: Bevacizumab; Device: NovoTTF-l00A; Other: Quality of Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab will be administered intravenously on days 1 and 15 of each 28 day cycle. The dose of bevacizumab will be 10 mg/kg of actual body weight.
  Other Names: Avastin; anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF
Device: NovoTTF-l00A — NovoTTF-100A will be worn continuously.
  Other Names: electric field therapy
Other: Quality of Life Assessment — Functional Assessment of Cancer Therapy including Brain Tumor module (FACT-Br) questionnaire
  Other Names: FACT-Br questionnaire

SUMMARY:
NovoTTF-100A is a device and Bevacizumab is a study drug that have both been approved by the FDA (Food and Drug Administration) for use as monotherapy in treating glioblastoma multiforme. The NovoTTF-l00A is a portable battery operated device which produces TTFields within the human body using surface electrodes (transducer arrays). Intermediate frequency electric fields (TTFields) stunt the growth of tumor cells.

The purpose of this study is to determine the efficacy of the combination of Bevacizumab and NovoTTF-100A in Bevacizumab naive (meaning have never received bevacizumab before) patients with recurrent glioblastoma (GBM) as measured by 6-month progression free survival.

DETAILED DESCRIPTION:
This will be an open label Phase II trial in adults with recurrent glioblastoma (GBM). The NovoTTF-100A treatment and Bevacizumab will be administered on an outpatient basis; NovoTTF-100A treatment will be initiated in the outpatient clinic.

PRIMARY OBJECTIVES:

I. To determine the efficacy of the combination of bevacizumab and NovoTTF-100A in bevacizumab-naive patients with recurrent glioblastoma (GBM) as measured by 6-month progression-free survival (PFS6).

SECONDARY OBJECTIVES:

I. To assess safety and tolerability of the combination of bevacizumab and Novo-TTF-100A in this patient population.

II. To evaluate overall survival in this population. III. To determine objective response rate (ORR) by modified Revised Assessment in Neuro-Oncology (RANO) criteria in this population.

IV. To assess time-to-progression in this population. V. To assess neurocognitive function (NCF) and quality of life (QOL) in this population.

OUTLINE:

Patients receive bevacizumab intravenously (IV) on days 1 and 15. Patients also undergo electric field therapy with NovoTTF-100A for at least 18 hours daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed glioblastoma or other grade IV malignant glioma (i.e. gliosarcoma, small cell glioblastoma, etc.), recurrent after prior external-beam fractionated radiotherapy and temozolomide chemotherapy.
* Patients with up to two prior recurrences are allowed.
* Karnofsky performance status ≥70.
* Patients must have the following laboratory values:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin (Hgb) > 9 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * ALT and AST ≤ 3.0 x ULN
  * Serum creatinine ≤ 1.5 x ULN
  * Blood coagulation parameters: INR ≤ 1.5
* Minimum interval since completion of radiation treatment is 12 weeks
* Minimum interval since last drug therapy:

  * 3 weeks since last non-cytotoxic therapy
  * 3 weeks must have elapsed since the completion of a non-nitrosourea-containing chemotherapy regimen
  * 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. The effects of bevacizumab on developing fetus or nursing infant are not known. Female patients of child-bearing potential must have a negative pregnancy test.
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission. Patients with other prior malignancies must be disease-free for ≥ three years.
* Patients must be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment and/or for at least 5 days before starting treatment.

Exclusion Criteria:

* Patients who have had previous treatment with bevacizumab, and or NovoTTF 100A system.
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias
  * Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)
  * Uncontrolled hypertension (defined by a systolic blood pressure (SBP) ≥ 160 mm Hg or diastolic blood pressure (DBP) ≥ 100 mm Hg while on anti-hypertensive medications)
* Patients with cirrhosis, or active viral or nonviral hepatitis.
* Implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain or documented clinically significant arrhythmias.
* Infra-tentorial tumor
* Evidence of increased intracranial pressure (clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* Known sensitivity to conductive hydrogels
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding women
* Patients unwilling or unable to comply with the protocol
* Patients with leptomeningeal disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09-18 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and NovoTTF-100A
Started | 25
Completed | 23
Not Completed | 2
Not completed — Screen failure | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants]
  10-19 years | 1
  20-29 years | 0
  30-39 years | 1
  40-49 years | 2
  50-59 years | 5
  60-69 years | 8
  70-79 years | 1
  unknown | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With 6-month Progression-free Survival (PFS6)
Description: Efficacy of therapy as measured by percent of participants with (PFS6). This trial will be considered successful if at least 20% of participants achieve PFS at 6 months. Disease progression is defined by RANO criteria. In cases where the RANO criteria cannot be applied, progression should be based on unequivocal evidence of progressive disease sufficient to require a change in therapy. The Modified RANO criteria are a set of guidelines for evaluating treatment response clinical trials. Modified RANO Response Criteria include levels of response including Complete Response (CR), Partial Response (PR), Minor Response (MR), Stable Disease (SD), or Progressive Disease.
Time Frame: 6 months
Population: Participants eligible for analysis (completed study)
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 23
percent of participants | 33 [9 to 60]

2. Secondary Outcome: Objective Response Rate (ORR) Based on RANO Criteria
Description: ORR as defined by the modified Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: 30 days after treatment completion through study completion, an average of 5 years, 9 months
Population: Only 16 of the 25 participants were analyzed because 9 participants were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 16
Participants
  Complete Response | 1
  Partial Response | 3
  Stable Disease | 6
  Progressive Disease | 6

3. Secondary Outcome: Number of Participants Experiencing Grade 3/4 Toxicities Related to Therapy Combination Per by CTCAE Version 4.0.
Description: Number of participants experiencing grade 3 or 4 toxicities related to therapy combination per by CTCAE version 4.0.
Time Frame: 5 years, 9 months
Population: All participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 25
Participants | 2

4. Secondary Outcome: Median Overall Survival
Description: Median overall survival (OS) in months
Time Frame: 30 days after treatment completion (Treatment continued until disease progression in the brain, death, or unacceptable side effects to patient)
Population: Participants eligible for analysis (completed study)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 23
months | 10.5 [8.2 to 14.9]

5. Secondary Outcome: Median Time-to-progression
Description: Median time to progression by Kaplan Meier methodology. Disease progression is defined by RANO criteria. In cases where the RANO criteria cannot be applied, progression should be based on unequivocal evidence of progressive disease sufficient to require a change in therapy. The Modified RANO criteria are a set of guidelines for evaluating treatment response clinical trials. Modified RANO Response Criteria include levels of response including Complete Response (CR), Partial Response (PR), Minor Response (MR), Stable Disease (SD), or Progressive Disease.
Time Frame: as for outcome 4
Population: Participants eligible for analysis (completed study)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 23
months | 4.1 [3.6 to 9.5]

6. Secondary Outcome: Time to Reliable Change in Neurocognitive Function (NCF)
Description: Time to reliable change in NCF by Kaplan Meier methodology. Memory, verbal fluency, visual-motor speed, executive function and motor dexterity tests will be administered. NCF testing involves standardized psychometric instruments that are sensitive to the neurotoxic effects of cancer treatment in brain tumor clinical trials.
Time Frame: as for outcome 4
Population: Only 2 participants reached reliable NCF change.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 2
months | 1.9 [0.14 to 3.7]

7. Secondary Outcome: Change From Baseline in Quality of Life (QOL) as Measured by FACT-BR Score
Description: Functional Assessment of Cancer Therapy including Brain Tumor module (FACT-Br) is a 54-item questionnaire that has four areas of cumulative measurements (physical well-being, social/family well-being, emotional well-being and functional well-being) with a scale of 0-4. The FACT-Br total score ranges between 0 and 76. The higher the score, the better the quality of life.
Time Frame: Baseline, 30 days after treatment completion (Treatment continued until disease progression in the brain, death, or unacceptable side effects to patient)
Population: Only 5 participants had QOL change from baseline.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 5
scores on a scale | 6 [-2 to 7]

8. Secondary Outcome: Percent of Participants With 12-month Progression-free Survival
Description: Efficacy of therapy as measured by percent of participants with 12-month PFS. Disease progression is defined by modified RANO criteria. In cases where the modified RANO criteria cannot be applied, progression should be based on unequivocal evidence of progressive disease sufficient to require a change in therapy. The Modified RANO criteria are a set of guidelines for evaluating treatment response clinical trials. Modified RANO Response Criteria include levels of response including Complete Response (CR), Partial Response (PR), Minor Response (MR), Stable Disease (SD), or Progressive Disease.
Time Frame: 12 months
Population: Participants eligible for analysis (completed study)
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Bevacizumab and NovoTTF-100A
Number analyzed (Participants) | 23
percent of participants | 19 [8 to 46]

ADVERSE EVENTS:
Time Frame: 5 years, 9 months
Arm/Group | Bevacizumab and NovoTTF-100A
All-Cause Mortality (participants affected / at risk) | 21/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and NovoTTF-100A (N=25)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (3)
Stroke (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and NovoTTF-100A (N=25)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Mucostis oral (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 8 (9)
Fatigue (General disorders) | 9 (12)
Gaid disturbance (General disorders) | 3 (3)
Irritability (General disorders) | 2 (3)
Pain (General disorders) | 2 (3)
Bronchial infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Alanine amiotransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (5)
Memory imparement (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 10 (24)
Throboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT01894061/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT01894061/ICF_001.pdf